CLINICAL TRIAL: NCT04772742
Title: Interventional, Randomized, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of Eptinezumab for the Preventive Treatment of Migraine in Patients With a Dual Diagnosis of Migraine and Medication Overuse Headache
Brief Title: Eptinezumab in Adults With Migraine and Medication Overuse Headache
Acronym: Sunlight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19139A
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Migraine; Medication Overuse Headache
MeSH Terms: conditions — Migraine Disorders; Headache Disorders, Secondary | interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eptinezumab (Experimental): Double-Blind Treatment Phase (at baseline): 100 mg eptinezumab by IV infusion
  Open-Label Treatment Phase (at week 12): 100 mg eptinezumab by IV infusion
  Interventions: Drug: Eptinezumab
- Placebo (Placebo Comparator): Double-Blind Treatment Phase (at baseline): Placebo by IV infusion
  Open-Label Treatment Phase (at week 12): 100 mg eptinezumab by IV infusion
  Interventions: Drug: Placebo; Drug: Eptinezumab

INTERVENTIONS:
Drug: Placebo — Placebo - solution for infusion
  Arms: Placebo
Drug: Eptinezumab — Eptinezumab - 100 mg, solution for infusion
  Other Names: Lu AG09221

SUMMARY:
This study evaluates the efficacy of eptinezumab to prevent migraine and headache in patients with the combined diagnosis of migraine and medication overuse headache

DETAILED DESCRIPTION:
Patients planned for randomization: 91 patients in the eptinezumab 100 mg group and 91 patients in the placebo group.

The total study duration from the Screening Visit to the Safety Follow-up Visit is approximately 36 weeks and includes a Screening Period (28-30 days), a Placebo-controlled Period (12 weeks), an Open-Label Period (12 weeks) and a Safety Follow-up Period (8 weeks). Patient will receive investigational medicinal product (IMP) at the Baseline Visit with either eptinezumab or placebo by IV infusion and at week 12 visit.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of migraine as defined by International Headache Society (IHS) International Classification of Headache Disorders (ICHD)-3 guidelines confirmed at the Screening Visit with a history of migraine onset of at least 12 months prior to the Screening Visit.
* The patient has ≥8 migraine days per month for each month on average within the past 3 months prior to the Screening Visit.
* The patient has a diagnosis of medication overuse headache (MOH) as defined by IHS ICHD-3 guidelines.
* The patient has headache on ≥15 days/month for each month within the past 3 months prior to the Screening Visit.
* The patient has regular overuse of one or more drugs that can be taken for acute and/or symptomatic treatment of headache, for >3 months.
* The patient has ≥15 to ≤26 headache days, of which ≥8 days were assessed as migraine days during the Screening Period, based on prospectively collected information in the eDiary.
* The patient overuses drugs that can be taken for acute and/or symptomatic treatment of headache during the Screening Period, based on prospectively collected information in the eDiary.
* The patient has demonstrated compliance with the Headache eDiary by entry of data for at least 24 of the 28 days of the Screening Period.
* The patient has had an onset of migraine at <50 years of age

Exclusion Criteria:

* The patient has experienced failure on a previous treatment targeting the calcitonin gene-related peptide (CGRP) pathway.
* The patient has confounding and clinically significant pain syndromes, (for example, fibromyalgia, chronic low back pain, complex regional pain syndrome).
* The patient has a diagnosis of acute or active temporomandibular disorder.
* The patient has a history or diagnosis of chronic tension-type headache, hypnic headache, cluster headache, hemicrania continua, new daily persistent headache, or unusual migraine subtypes such as hemiplegic migraine (sporadic and familial), recurrent painful ophthalmoplegic neuropathy, migraine with brainstem aura and migraine with neurological accompaniments that are not typical of migraine aura (diplopia, altered consciousness, or long duration).
* Patients with a lifetime history of psychosis, bipolar mania, or dementia are excluded. Patients with other psychiatric conditions whose symptoms are not controlled or who have not been adequately treated for a minimum of 6 months prior to screening are also excluded.
* The patient has a history of clinically significant cardiovascular disease, including uncontrolled hypertension, vascular ischaemia or thromboembolic events (for example, cerebrovascular accident, deep vein thrombosis, or pulmonary embolism).

Other in- and exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the number of monthly migraine days (MMDs) | Weeks 1-12

SECONDARY OUTCOMES:
Change from baseline in MMDs with use of acute medication | Weeks 1-12
Response: ≥50% reduction from baseline in MMDs | Weeks 1-12
Migraine rate on the day after dosing | At Day 1
Response: ≥75% reduction from baseline in MMDs | Weeks 1-4
Change from baseline in the number of monthly headache days (MHDs) | Weeks 1-12
Response: ≥75% reduction from baseline in MMDs | Weeks 1-12
Response: ≥75% reduction from baseline in MHDs | Weeks 1-12
Response: ≥75% reduction from baseline in MHDs | Weeks 1-4
Change from baseline in the number of MHDs with use of acute medication | Weeks 1-12
Change from baseline in rate of migraines with severe pain intensity | Weeks 1-12
Change from baseline in rate of headaches with severe pain intensity | Weeks 1-12
Patient Global Impression of Change (PGIC) score | At Week 12
Most Bothersome Symptom (MBS) (score as measured relative to Screening) | At Week 12
Change from baseline to Week 12 in the Headache Impact Test (HIT-6) score | Baseline to Week 12
Change from baseline to Week 12 in the Migraine-Specific Quality of Life (MSQ v2.1) sub-scores (Role Function-Restrictive, Role Function-Preventive, Emotional Function) | Baseline to Week 12
Change from baseline to Week 12 in the Health-Related Quality of Life (EQ-5D-5L) Visual Analogue Scale (VAS) score | Baseline to Week 12
Health Care Resources Utilization (HCRU) | Baseline to Week 12
  Migraine-specific healthcare resource utilization information will be collected in terms of outpatient health care professional visits, emergency room visits, hospital admissions, as well as duration of hospital stays.
Change from baseline to Week 12 in the Work Productivity and Activity impairment Questionnaire: Migraine (WPAI:M) sub-scores (Absenteeism, Presenteeism, Work productivity loss, Activity impairment) | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (40):
- China (26):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Beijing Chaoyang Hospital Capital Medical University, Beijing
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Peking University First Hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Beijing
  - The First Hospital of Jilin University, Changchun
  - The Second Hospital of Jilin University, Changchun
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Mianyang Central Hospital, Mianyang
  - Jiangxi Pingxiang People's Hospital, Pingxiang
  - People's Hospital of Rizhao, Rizhao
  - Shengjing Hospital of China Medical University, Shenyang
  - General Hospital of Northern Theater Command, Shenyang
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen
  - Shanxi Provincial People Hospital, Taiyuan
  - The 2nd Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - People's Hospital of Zhengzhou, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- Georgia (2):
  - Pineo Medical Ecosystem, Tbilisi
  - Aversi Clinic LTD, Tbilisi
- South Korea (3):
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
- Spain (6):
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Taiwan (3):
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Yu S, Zhou J, Luo G, Xiao Z, Ettrup A, Jansson G, Florea I, Ranc K, Pozo-Rosich P. Efficacy and safety of eptinezumab in patients with chronic migraine and medication-overuse headache: a randomized, double-blind, placebo-controlled study. BMC Neurol. 2023 Dec 15;23(1):441. doi: 10.1186/s12883-023-03477-z. PMID 38102535